CLINICAL TRIAL: NCT02177916
Title: "A Comparison of 2 Different Methods of Patient Education to Determine Knowledge Acquisition in Patients Preparing to Undergo Lung Transplantation"
Brief Title: Patient Education Study to Determine Knowledge Acquisition in Patients Preparing to Undergo Lung Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampa General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: TGH0004
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Lung Transplantation
Keywords: lung transplantation
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional teaching (Experimental)
  Interventions: Other: Education
- DVD (Experimental)
  Interventions: Other: Education

INTERVENTIONS:
Other: Education

SUMMARY:
The Lung Transplant Team at Tampa General Hospital has identified a need to improve both the quality and quantity of the education that is provided to patients listed for lung transplantation. We propose to change the method and timing of our transplant patient education. The objective of this prospective data collection will be to collect and analyze pre and post test scores of patients when patient education is provided via compact disc as compared to individualized teaching.

ELIGIBILITY:
Inclusion Criteria:

* Age- 18-75

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of patient education when provided via compact disk as compared to individualized teaching as assessed by pre and post test scores. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rolfe, MD, Principal Investigator — Tampa General Hospital
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States